CLINICAL TRIAL: NCT07240402
Title: Comparative Study of Morphine and Dexmedetomidine as Adjuvants to Bupivacaine in Ultrasound-Guided Adductor Canal Block for Postoperative Analgesia After Knee Surgeries
Brief Title: Compare Morphine and Dexmedetomidine as Adjuvants to Bupivacaine in Ultrasound-guided ACB for Postoperative Analgesia After Knee Surgeries
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ashraf Abd El-Nasser Abd El-Hamid, Ashraf Elrewany, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KafrelsheikhU
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Analgesia; Morphine and Dexmedetomidine
Keywords: Adductor Canal Block
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group D (Experimental): Patients will receive ACB using 20 ml of bupivacaine 0.25%+ 0.5 µg/kg dexmedetomidine.
  Interventions: Drug: Adductor Canal Block (ACB) Only
- Group M (Experimental): Patients will receive ACB using 20 ml of bupivacaine 0.25%
  +0.1 mg/kg morphine.
  Interventions: Drug: Adductor Canal Block (ACB) Only
- Group C (Experimental): Patients will receive ACB using 20 ml of bupivacaine 0.25% alone as a control group.
  Interventions: Drug: Adductor Canal Block (ACB) Only

INTERVENTIONS:
Drug: Adductor Canal Block (ACB) Only — This study aims to compare morphine and dexmedetomidine as adjuvants to bupivacaine in ultrasound-guided ACB for postoperative analgesia after knee surgeries. Primary outcome:
  • Time to first rescue analgesia .
  Secondary outcomes:
  * Total opioid consumption in 24 hours postoperatively.
  * Degree of pain using visual analogue scale (VAS).
  * Degree of patient satisfaction.
  * Incidence of complication A) Related to block Nerve Injury Vascular Puncture Hematoma B) Related to drug Local Anesthetic Systemic Toxicity (LAST)
  Other Names: adductor canal block

SUMMARY:
This study aims to compare morphine and dexmedetomidine as adjuvants to bupivacaine in ultrasound-guided ACB for postoperative analgesia after knee surgeries

DETAILED DESCRIPTION:
Knee surgeries are frequently performed operations that can lead to intense pain after the procedure (1). Early mobilization following knee surgery is associated with improved functional outcomes and a reduction in postoperative complications. As a result, achieving effective pain relief while preserving motor function is a primary goal in postoperative care for knee procedures (2).

A variety of strategies are employed for managing postoperative pain, including systemic opioid administration, epidural anesthesia, peripheral nerve blocks, and local infiltration of anesthetics (3).

However, systemic opioids are linked to several undesirable side effects such as nausea, vomiting, itching, sedation, and respiratory depression, which may hinder rehabilitation.

Similarly, epidural analgesia often results in complications like hypotension, urinary retention, and pruritus. The use of long-acting intrathecal opioids has also been associated with adverse events including bilateral motor blockade, tremors, and hypotension. Due to these issues, the reliance on systemic and intrathecal methods for postoperative pain control has been declining (4).

The adductor canal block (ACB), which targets the Hunter's canal, anesthetizes the saphenous and vastus medialis nerves, along with partial coverage of other sensory nerves like the femoral nerve, medial cutaneous nerve, and branches of the obturator nerve as they traverse the distal canal (5). ACB is largely considered a sensory block, affecting only the motor nerve to the vastus medialis, making it advantageous in preserving quadriceps strength during recovery (6, 7). Bupivacaine, a widely used long-acting amide local anesthetic, is frequently employed in peripheral nerve blocks such as the ACB due to its favorable pharmacokinetics.

Nonetheless, its analgesic duration may be insufficient for managing postoperative pain in surgeries with high nociceptive intensity (8). To extend its efficacy and enhance analgesic quality, several adjunctive agents have been explored, including opioids and α2-adrenergic agonists (9).

Morphine, a traditional opioid analgesic, acts on μ-opioid receptors to prolong analgesia and reduce local anesthetic requirements. Despite its effectiveness, its use is limited by opioid-related adverse effects like nausea, vomiting, pruritus, and respiratory depression. Furthermore, some studies report that morphine may not significantly improve postoperative pain control or functional recovery after knee surgery (10-12).

Dexmedetomidine, a highly selective α2-adrenergic receptor agonist, has been increasingly studied as an adjuvant in peripheral nerve blocks. When administered

perineurally, it has demonstrated potential to accelerate onset, prolong analgesia, reduce postoperative pain intensity, and minimize systemic opioid use, all while producing fewer systemic side effects (13). Its peripheral analgesic properties are thought to result from direct binding to α2-receptors at the nerve site (14).

Currently, there is limited research directly comparing the efficacy of morphine versus dexmedetomidine as adjuvants to bupivacaine in ultrasound-guided ACB for postoperative analgesia following knee surgeries.

ELIGIBILITY:
Inclusion criteria:

* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Body mass index (BMI) of 20-35 kg/m2.
* Undergoing knee surgeries under spinal anesthesia.

Exclusion criteria:

* Any known allergy or contraindication to local anesthetic.
* History of substance abuse.
* Decompansated cardiac, pulmonary, hepatic, renal disease.
* Obese patients with BMI>35kg/m2.
* Pregnant and lactating mothers.
* Coagulopathies.
* Local skin infections at the site of injection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: | 24 hours postoperatively.
  • Time to first rescue analgesia .

IPD SHARING:
Plan to Share IPD: No